CLINICAL TRIAL: NCT02697786
Title: The Impact of Intraoperative Microemboli Load on Postoperative Brain Injury in Patients Undergoing Aortic Valve Replacement Preformed With Two Different Surgical Approaches
Brief Title: Neuromonitoring in Patients During Aortic Valve Replacement
Acronym: IMLPBIAVR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Marija Bozhinovska (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Sponsor-Investigator, Marija Bozhinovska, MD, MSc, Spec., University Medical Centre Ljubljana
Organization: University Medical Centre Ljubljana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ARRS-RPROJ - J R- 2014- 191
Record Dates: First submitted 2016-01-25; First posted 2016-03-03 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Brain Injury
Keywords: Aortic valve surgery
MeSH Terms: conditions — Brain Injuries | interventions — Ultrasonography, Doppler, Transcranial

ARMS (2):
- AVR preformed with full sternotomy (Active Comparator): 30 patients, 7 days before and after surgery mini mental test and measurement of visual evoked cerebral blood flow response (VEFR) will be done.
  Transcranial doppler measurements 1. beginning of the surgery, 2.after sternotomy, 3.during aortic cannulation,4.during CPB,5. during de-airing, 6. opening of the clamp on the aorta, 7. after CPB removal before chest closure. Prolonged de airing if needed
  Interventions: Device: Transcranial doppler
- AVR preformed with minimal invasive sternotomy (Experimental): 30 patients, 7 days before and after surgery mini mental test and measurement of visual evoked cerebral blood flow response (VEFR) will be done.
  Transcranial doppler measurements 1. beginning of the surgery, 2.after sternotomy, 3.during aortic cannulation,4.during CPB,5. during de-airing, 6. opening of the clamp on the aorta, 7. after CPB removal before chest closure. Prolonged de airing if needed
  Interventions: Device: Transcranial doppler

INTERVENTIONS:
Device: Transcranial doppler — Prolonged de airing to decrease the number of MES

SUMMARY:
Postoperative brain damage and neuropsychological disorders have been observed in 30 - 80 % of patients after heart surgery with the use of cardiopulmonary bypass (CPB).They can persist up to a year after cardiac surgery and are associated with increased hospital mortality and prolonged intrahospital stay.

Hypoperfusion,hyperthermia,atrial fibrillation,genetic predisposition and systemic inflammatory response associated with CPB have been identified as pathophysiological mechanisms.However, some authors consider cerebral embolisation to be the prevalent mechanism of intraoperative brain injury after cardiac surgery,as gaseous or solid cerebral emboli can cause ischemia, inflammation and edema,consequently causing cerebral infarctions usually resulting with stroke,coma,encephalopathy, delirium and cognitive decline. Additionally,they may impair cerebrovascular reactivity (CVR).

Aortic valve replacement (AVR) preformed by full sternotomy is the standard approach in the treatment of aortic valve disease. Minimally invasive (MIS) aortic valve replacement has been shown to reduce postoperative mortality, morbidity, and pain while providing faster recovery, a shorter hospital stay, and better cosmetic results. However, due to technically more demanding procedure, MIS may lead to prolonged CPB time and incomplete de-airing of the heart with an increased risk for cerebral gas embolization. Therefore, the choice of MIS might bear an augmented risk for brain injury.

Transcranial Doppler (TCD) enables real time detection of intraoperative emboli in the cerebral arteries seen as microembolic signals (MES), and is an essential neuromonitoring tool. Several studies demonstrated correlation between the number of MES and the occurrence as well as severity of postoperative neurological complications. However, the factors contributing to brain injury have not been elucidated in those studies. The investigators speculate that impairment of CVR is an important mechanism that persists and prolongs the duration of brain injury into postoperative period.

The aim of the study is to compare two surgical approaches used for AVR, with focus on the number of MES and their impact on levels of protein S100B (marker of brain tissue damage),postoperative CVR and cognitive function With the results,the investigators aim to help surgeons in selecting the appropriate technique for AVR in individual participants,as well as to clarify the effect of aortic valve surgery on the brain.

DETAILED DESCRIPTION:
Patients undergoing for aortic valve replacement will be enrolled in the study after giving the signed informed consent and will be divided in two groups depending on the type of the surgical technique. Either full sternotomy (FS) or minimal invasive sternotomy (MIS) will be performed, both with the use of cardio-pulmonary bypass (CPB).One week before and one week after the surgery patients will undergo mini mental test and measurement of visually evoked cerebral blood flow velocity response (VEFR).Levels of S100B, interleukin (IL) 1, IL 6, IL 8, IL 10 and microparticles will be determined before induction of anesthesia,as well as 6 h, 24 h, 48 h and 7 days after CPB.Each patient will have invasive and non invasive monitoring that will include near infrared spectroscopy (NIRS), bispectral index (BIS) and TCD during surgery.MES will be detected using TCD at the following time-points: beginning of surgery, after sternotomy, during aortic cannulation, during CPB, during de-airing, opening of the clamp on the aorta and after CBP removal before chest closure.All of this data will be documented as well as the demographic characteristics of patients, their preoperative medical status, and intraoperative data (duration of surgery, duration of CPB, hemodynamic parameters, inotropic/vasoactive support,blood and blood components); duration of mechanical ventilation in intensive care unit (ICU), duration of ICU stay, 30-day mortality and morbidity, as well as postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Isolated aortic valve stenosis as well as asymptomatic patients with depressed systolic function
* Symptomatic patients with normal or depressed left ventricular function
* Patients with American Society of Anesthesiologist (ASA) physical status classification 2 or 3

Exclusion Criteria:

* History of brain stroke
* EF less than 20%
* History of alcohol abuse
* Epilepsy of history of psychiatric illness and antipsychotic drugs
* Patients with stenosis on carotid arteries
* Patients with preformed surgery or already stented carotid arteries
* Patients with poor or absent acoustic temporal window
* Diagnosed dementia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Detection of the intraoperative microembolic signals during minimal invasive sternotomy compared to full sternotomy with TCD during aortic valve surgery | Intraoperative detection:Beginning of surgery, after sternotomy, during aortic cannulation, during CPB, during de-aeration, opening of the clamp on the aorta and after CBP removal before chest closure.
Detection of S100B serum protein, marker of brain tissue damage | Before induction of anesthesia, 6 h , 24 h, 48h and 7 days after CPB
Detection of serum interleukin IL-1, IL-6,IL-8,Il-10 and Microparticles | Before induction of anesthesia, 6 h , 24 h, 48h and 7 days after CPB

SECONDARY OUTCOMES:
Assessment of cerebrovascular reactivity using visually evoked cerebral blood flow velocity response (VEFR) measurements | 7 days before and 7 days after surgery
Assessment of neurologic and cognitive function in patients undergoing AVR | 7 days before and 7 days after surgery

OTHER OUTCOMES:
Length of ICU stay | Post operative period, an expected average of 2 days
Requirement for inotropic and vasoactive therapy | 1)After induction of anesthesia, 2)at the end of CPB ,3) postoperative period
Duration of mechanical ventilation | postoperative period, an expected average 2 days
30 days mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Maja Sostaric, MD, PhD, Study Director — University Medical Centre Ljubljana; Matej Podbregar, MD, PhD, Study Director — University Medical Centre Ljubljana; Tomislav Klokocovnik, MD,PhD, Study Director — University Medical Centre Ljubljana; Borut Gersak, MD, PhD, Study Director — University Medical Centre Ljubljana; Marija Bozhinovska, MD, MSc, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Clinical center, Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bozhinovska M, Jenko M, Stupica GT, Klokocovnik T, Ksela J, Jelenc M, Podbregar M, Fabjan A, Sostaric M. Cerebral microemboli in mini-sternotomy compared to mini- thoracotomy for aortic valve replacement: a cross sectional cohort study. J Cardiothorac Surg. 2021 May 24;16(1):142. doi: 10.1186/s13019-021-01509-8. PMID 34030698